CLINICAL TRIAL: NCT04548895
Title: Non-invasive Biometric Monitoring for the Prevention of COVID-19 Transmission and Deaths in Nursing Homes
Brief Title: Non-invasive Biometric Monitoring in Nursing Homes to Fight COVID-19
Status: Completed | Type: Observational
Sponsor: Health Stream Analytics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HSA-001
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Community-Acquired Respiratory Tract Infection
Keywords: COVID-19; wearables; biometric data
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: None Retained — Nasal swabs will be taken at five time points to test for virus presence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LTCF residents and involved health practitioners: The intervention will take place in nursing homes, assisted living facilities and long-term care facilities (LTCF) in the United States (henceforth collectively referred to as "LTCF").
  Staff who work in the participating LTCF ≥ 20 hours/week and who have direct contact with the residents are also eligible to participate and to employ the biometric monitoring equipment in their private residences.
  Interventions: Device: Observational measurement of biometric data. No change to health care provided.

INTERVENTIONS:
Device: Observational measurement of biometric data. No change to health care provided. — Emfit devices will be installed once after enrollment under each participant's mattress and left to record automatically without further intervention. The participants will wear their Biostrap wristbands consistently, ideally 24 hours a day, 7 days a week, for 2 months.
  A virus panel will be upon enrollment (baseline) and then every two weeks (± 3 days, or on the closest convenient sampling day if the LTCF is testing all residents on the same day) for a maximum of 5 times during the two-month period. Using polymerase chain reaction or next generation sequencing, the virus panel will detect COVID-19 and 12 other common respiratory viruses that may cause similar symptoms and similar biometric signatures. These include influenza A and B, parainfluenza types 1 through 4, respiratory syncytial virus, non-COVID coronavirus, rhinovirus, adenovirus, bocavirus and metapneumovirus.

SUMMARY:
Solving the problem of detecting asymptomatic carriers who can transmit infection is key to protecting vulnerable residents of nursing homes and assisted living facilities, to protecting frontline workers who care for them, and to facilitating return to work (including return of nurses and medical assistants).

The wearable biometric technology, if widely disseminated among vulnerable populations and the community-at-large, will help avoid the ravages of seasonal flu and other contagious illnesses, and the society will be better prepared for future waves of COVID-19 or other pandemics. Even if a vaccine is developed, due to immune senescence and immunocompromise, elderly people and those with chronic medical conditions may not be well protected by it. Continuous biomonitoring provides another layer of protection for them.

DETAILED DESCRIPTION:
1. Building the algorithm for early, pre-symptomatic DETECTION OF RESPIRATORY VIRAL INFECTION and for predicting eventual DETERIORATION.
2. Create an APP that AUTOMATES these algorithms and clearly REPORTS ACTIONABLE RESULTS to users, i.e., to medical professionals and citizens-at-large in near-real time. If alerted to a possible - and likely still asymptomatic - COVID-19 infection, they can self-isolate or be quarantined, get confirmatory COVID-19 testing done promptly, limit transmission to others, and stay safe knowing that if they are likely to deteriorate, the algorithm will alert the participants and their caregivers to the need to obtain medical attention promptly.

ELIGIBILITY:
Inclusion Criteria:

* Residents and staff members of U.S. LTCFs where COVID-19 transmission is actively occurring. The LTCF medical director must agree to enroll the LTCF, and each participant must have the capacity to agree and sign consent.

Exclusion Criteria:

* Current atrial fibrillation.

  * NB: Paroxysmal atrial fibrillation is permitted if the participant is in atrial fibrillation less than 50% of the day on most days.
* Pacemaker in place.
* Known active infection other than COVID-19.
* Dementia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents and staff members of U.S. LTCFs where COVID-19 transmission is actively occurring. The LTCF medical director must agree to enroll the LTCF, and each participant must have the capacity to agree and sign consent.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Proportion of quality signals obtained out of all monitoring time for each device | 8 weeks from first enrollment
  Feasibility assessment
Predictive characteristics of the algorithm for respiratory tract infection | 2 months
  Algorithm development, sensitivity, specificity, positive and negative predictive value at different lead times ahead of symptom onset

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Frasch, Study Chair — Health Stream Analytics, LLC
Locations (1):
- Avalon Health & Rehabilitation Center, Pasco, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: At least 55,000 or more than 40% of currently over 120,000 deaths from COVID-19 were residents and workers at nursing homes and other long-term care facilities for older adults in the United States. — https://www.nytimes.com/interactive/2020/us/coronavirus-nursing-homes.html